CLINICAL TRIAL: NCT00863070
Title: Biomechanical Assessment of Level Gait in Patient's Status Post Bladder Exstrophy
Acronym: Gait
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-003
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Bladder Exstrophy
Keywords: Bladder exstrophy; Abnormal gait; anatomy; urinary bladder disease; urogenital abnormalities
MeSH Terms: conditions — Bladder Exstrophy; Mobility Limitation; Urinary Bladder Diseases; Urogenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bladder Exstrophy Patients: Patients who receive follow-up care at Connecticut CMC urology clinic for bladder exstrophy.

SUMMARY:
The purpose of this study is to determine whether patients who have undergone exstrophy closure may be at risk for long-term orthopedic issues manifest by gait abnormalities. This study is a descriptive analysis of the study cohort's gait patterns and pelvic structure.

Specific Aim 1: to determine whether patients with classic bladder exstrophy who underwent closure demonstrate gait abnormalities.

Hypothesis 1: Patients undergoing closure of bladder exstrophy (with or without pelvic osteotomy) demonstrate gait abnormalities compared with a reference population.

Hypothesis 2: Patients undergoing closure of bladder exstrophy (with or without pelvic osteotomy) will have below normal functional survey scores.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was seen at CCMC for bladder exstrophy between January 2002 and December 2010.
2. Subject is four years of age or older at time of enrollment.
3. Subject has the ability to walk.
4. Subject has not had gait testing performed.
5. Subject provides Informed Consent and HIPAA Authorization.

Exclusion Criteria:

1. Subject was not seen at CCMC for bladder exstrophy between January 2002 and December 2010.
2. Subject under four years of age at time of enrollment.
3. Subject does not have the ability to walk.
4. Subject had prior gait testing performed.
5. Subject not willing to provide Informed Consent and HIPAA Authorization.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bladder exstrophy patients receiving follow-up services at Connecticutcmc Urology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Gait Testing and Analysis | 2 Weeks

SECONDARY OUTCOMES:
Demographic Data:age;GA at birth; Prenatal DX;closure age;Pelvic osteotomies;Perioperative and late complications;Successful initial closure;Continence; Additional surgeries w/age | 2 weeks
Pediatric Outcomes Data Collection Instrument (PODCI) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine W Herbst, M.Sc, Study Director — Connecticut Children's Medical Center
Locations (2):
- United States (2):
  - Center for Motion Analysis, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No